CLINICAL TRIAL: NCT04373941
Title: Granulocyte-Colony Stimulating Factor Adjunct Therapy for Biliary Atresia: Part II of a Prospective, Randomized Controlled, Multi-Institutional Trial
Brief Title: Part II: Granulocyte-Colony Stimulating Factor Adjunct Therapy for Biliary Atresia
Acronym: BA_GCSF2b
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holterman, Ai-Xuan, M.D. (Individual)
Collaborators: T Rose Clinical, Inc. (Unknown); Big Leap Research (Other); Prometheus USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HoltermanA
Record Dates: First submitted 2019-08-13; First posted 2020-05-05 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: GCSF or No-GCSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Kasai GCSF (Experimental): The Kasai GCSF group will receive the standard of care PLUS 3 consecutive daily doses of 10 ug/kg of GCSF to be administered subcutaneously by day 3 post Kasai surgery
  Interventions: Drug: Filgrastim
- Kasai no GCSF (No Intervention): The no GCSF group will not receive GCSF and receives the standard of care
- No Kasai GCSF (Experimental): The No Kasai GCSF group will receive the standard of care PLUS 3 consecutive daily doses of 10 ug/kg of GCSF to be administered subcutaneously once the diagnosis of BA is established
  Interventions: Drug: Filgrastim
- No Kasai No GCSF (No Intervention): The No Kasai No GCSF group will receive the standard of care and will not receive GCSF

INTERVENTIONS:
Drug: Filgrastim — G-CSF is a glycoprotein produced by monocytes, fibroblasts, and endothelial cells. Filgrastim is a human granulocyte colony stimulating factor (G-CSF) produced by recombinant DNA technology with NEUPOGEN® as the Amgen Inc. trademark for filgrastim. G-CSF regulates the production, proliferation and differentiation of neutrophils and hematopoietic stem cell precursors within the bone marrow leading to dose-dependent increase in circulating neutrophils and hematopoietic stem cells in the blood. It is indicated to reduce the incidence of infection in patients with severe neutropenia, for neutrophil recovery in neutropenic patients with bone marrow depletion, to mobilize hematopoietic progenitor stem cell for collection by leukapheresis in hematopoietic stem cell transplantation.
  Other Names: Neupogen, granulocyte colony stimulating factor
  Arms: Kasai GCSF; No Kasai GCSF

SUMMARY:
The Investigators propose to test the hypothesis that GCSF enhances the clinical outcome of biliary atresia in a multi-institutional Phase 2 trial to prospectively evaluate the safety and efficacy of GCSF in each of the 2 groups of newly diagnosed BA patients: KBA (i.e., Kasai-operated) or NoK (i.e., patients who did not undergo Kasai surgery). Subjects who participate in the trial will be followed for 2 years.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-institutional trial in KBA and NoK subjects to be conducted under a Food and Drug Administration approved Investigational New Drug application.

The KBA group is composed of just operated Kasai patients with intraoperative liver biopsy-confirmed BA. Their clinical characteristics have been described in the previously completed Phase 1 study under CR00005169 (ie. inclusion and exclusion criteria as described below)

The NoK group will be composed of newly diagnosed BA patients, including the following:

* surgical patients in whom the Kasai was not performed for intraoperative technical reasons or due to advanced liver disease, who also have no option for rescue liver transplantation.
* Unoperated patients whose family refuses surgery or who are not operative candidates

Having met the same inclusion and exclusion criteria as the Kasai KBS group,

* eligible KBA subjects will be randomized to GCSF vs. no-GCSF at the 10 ug/kg/d dose to be given subcutaneously for 3 consecutive daily doses on the third day following the Kasai procedure.
* eligible NoK subjects will be randomized to GCSF vs. no-GCSF at the 10 ug/kg/d dose to be given subcutaneously for 3 consecutive daily doses on the third day following diagnostic liver biopsy.

ELIGIBILITY:
Inclusion criteria

1. preliminary work up for cholestasis suspected or inconclusive diagnosis of BA.
2. Serum Direct bilirubin > 2 mg/dl,GGT> 100 U/L
3. Male or female infants with a gestational age> 36 weeks
4. Admission weight > 2 kg
5. Age > 14 days - 180 days at diagnosis
6. For Kasai operated subjects, Type 3 or 4 anatomy of BA
7. For Kasai operated subjects, cholangiogram (if performed) diagnostic of BA
8. Liver biopsy supporting BA diagnosis

Exclusion criteria

1. Patients having access to liver transplantation for immediate liver failure
2. Prior Kasai patients
3. Major cardiac, renal, central nervous system (CNS) malformations
4. Intracranial hemorrhage
5. History of recent total parenteral nutrition (TPN) use within the last 2 weeks
6. Gl tract obstruction

   For Kasai-operated subjects: Type 1 or 2 biliary atresia anatomy
7. Current systemic infection
8. WBC > 20,000 cells/uL
9. Platelet count < 20,000 cells/uL or >1 million cells/uL
10. Concurrent respiratory, metabolic, neurological, cardiovascular, metabolic, and renal illness
11. Elevated serum creatinine > 1 mg/dL
12. Purpura fulminans or unexplained vascular thrombosis

Ages: 14 Days to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
GCSF Response on Bile flow (KBA) | 3 months
  For KBA subjects: Bile flow as measured by the percentage of subjects with total bilirubin< 2 mg/dL at 3 months post-Kasai.
GCSF Response on transplant-free survival (NoK) | 24 months
  For NoK subjects: Changes at 6, 12, 18 and 24 months-transplant free survival

SECONDARY OUTCOMES:
GCSF response on liver function and outcome (KBA) | 24 months
  KBA subjects: Pediatric end-stage liver disease (PELD) score at 6, 12, 18, and 24 months after GCSF treatment.
GCSF response on liver function and outcome (KBA) | 24 months
  KBA subjects: Percentage of patients with transplant-free survival at 6, 12, 18 and 24 months
GCSF response on liver function and outcome (KBA) | 24 months
  KBA subjects: Percentage of patients with cholangitis-free transplant-free survival at 6, 12, 18 and 24 months
GCSF response on liver function (NoK) | 24 months
  NoK subjects: Changes in Pediatric end-stage liver disease (PELD) score at 6, 12, 18, and 24 months after GCSF treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States
- Aga Khan University, Karachi, Pakistan
- Vietnam (2):
  - Nation Children's Hospital, Hanoi, Dong Da District
  - Children Hospital 1, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezerra JA, Wells RG, Mack CL, Karpen SJ, Hoofnagle JH, Doo E, Sokol RJ. Biliary Atresia: Clinical and Research Challenges for the Twenty-First Century. Hepatology. 2018 Sep;68(3):1163-1173. doi: 10.1002/hep.29905. PMID 29604222
- [Background] Chaudhuri J, Mitra S, Mukhopadhyay D, Chakraborty S, Chatterjee S. Granulocyte Colony-stimulating Factor for Preterms with Sepsis and Neutropenia: A Randomized Controlled Trial. J Clin Neonatol. 2012 Oct;1(4):202-6. doi: 10.4103/2249-4847.105993. PMID 24027727
- [Background] Shneider BL, Magee JC, Karpen SJ, Rand EB, Narkewicz MR, Bass LM, Schwarz K, Whitington PF, Bezerra JA, Kerkar N, Haber B, Rosenthal P, Turmelle YP, Molleston JP, Murray KF, Ng VL, Wang KS, Romero R, Squires RH, Arnon R, Sherker AH, Moore J, Ye W, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Total Serum Bilirubin within 3 Months of Hepatoportoenterostomy Predicts Short-Term Outcomes in Biliary Atresia. J Pediatr. 2016 Mar;170:211-7.e1-2. doi: 10.1016/j.jpeds.2015.11.058. Epub 2015 Dec 24. PMID 26725209
- [Background] Kedarisetty CK, Anand L, Bhardwaj A, Bhadoria AS, Kumar G, Vyas AK, David P, Trehanpati N, Rastogi A, Bihari C, Maiwall R, Garg HK, Vashishtha C, Kumar M, Bhatia V, Sarin SK. Combination of granulocyte colony-stimulating factor and erythropoietin improves outcomes of patients with decompensated cirrhosis. Gastroenterology. 2015 Jun;148(7):1362-70.e7. doi: 10.1053/j.gastro.2015.02.054. Epub 2015 Mar 4. PMID 25749502
- [Background] Fanna M, Masson G, Capito C, Girard M, Guerin F, Hermeziu B, Lachaux A, Roquelaure B, Gottrand F, Broue P, Dabadie A, Lamireau T, Jacquemin E, Chardot C. Management of Biliary Atresia in France 1986 to 2015: Long-term Results. J Pediatr Gastroenterol Nutr. 2019 Oct;69(4):416-424. doi: 10.1097/MPG.0000000000002446. PMID 31335841
- [Background] Verma N, Kaur A, Sharma R, Bhalla A, Sharma N, De A, Singh V. Outcomes after multiple courses of granulocyte colony-stimulating factor and growth hormone in decompensated cirrhosis: A randomized trial. Hepatology. 2018 Oct;68(4):1559-1573. doi: 10.1002/hep.29763. Epub 2018 Jul 25. PMID 29278428
- [Background] Spahr L, Lambert JF, Rubbia-Brandt L, Chalandon Y, Frossard JL, Giostra E, Hadengue A. Granulocyte-colony stimulating factor induces proliferation of hepatic progenitors in alcoholic steatohepatitis: a randomized trial. Hepatology. 2008 Jul;48(1):221-9. doi: 10.1002/hep.22317. PMID 18537187
- [Background] Korbling M, Freireich EJ. Twenty-five years of peripheral blood stem cell transplantation. Blood. 2011 Jun 16;117(24):6411-6. doi: 10.1182/blood-2010-12-322214. Epub 2011 Apr 1. PMID 21460243
- [Derived] Nguyen HPA, Ren J, Butler M, Li H, Qazi S, Sadiq K, Dao HT, Holterman A. Study protocol of Phase 2 open-label multicenter randomized controlled trial for granulocyte-colony stimulating factor (GCSF) in post-Kasai Type 3 biliary atresia. Pediatr Surg Int. 2022 Jul;38(7):1019-1030. doi: 10.1007/s00383-022-05115-0. Epub 2022 Apr 7. PMID 35391541